CLINICAL TRIAL: NCT03997110
Title: Rapid Palliation in Locally Advanced Cervical Cancer: A Phase III Randomized Trial
Brief Title: Palliative Radiation for Advanced Cervical Cancer
Acronym: RAPPAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Memorial Hospital (Other Government)
Collaborators: Tata Memorial Centre (Other)
Responsible Party: Principal Investigator, Supriya Sastri (chopra), Professor, Tata Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMH IRB 3157
Record Dates: First submitted 2019-04-09; First posted 2019-06-25 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Cervical Cancer
Keywords: Cervical Cancer; Palliative treatment; Radiation Therapy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Phase III, Randomized, Active Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A Or Control Arm- Long course palliative treatment. (Active Comparator): Week1: All the patients will receive external sitting of radiation treatment, first fraction of 10 Gy. Week4: All the patients will receive external sitting of radiation treatment, second fraction of 10 Gy. Week7: Patients who have almost complete clinical response will be evaluated for brachytherapy will receive the appropriate brachytherapy procedure depending on the tumor response to a dose of 6-8Gy x 2-3#.The patients who will be found unsuitable for brachytherapy will receive another sitting of external radiation, third fraction of 10 Gy. Week 12: After treatment completion response assessment will be done using following parameters: • Pain assessment using numerical pain rating scale on 0-10 • Vaginal bleeding- yes/ no • Vaginal discharge- yes/no • Analgesic use- WHO ladder and dosing • QOL QC30, QLQC15 Pall, QLQC Cervix 24 • Disease response • Acute toxicity
  Interventions: Radiation: Long course palliative treatment.
- Arm B or Experimental Arm-Short course palliative radiation. (Experimental): Week 1: Patients in the experimental arm will be treated with short course radiotherapy (25Gy/5#). The dose fractionation of 25 Gy in 5# over a week will be used. Week 4: Patients who have almost complete clinical response will be evaluated for brachytherapy will receive the appropriate brachytherapy procedure depending on the tumor response to a dose of 6-8Gy x 2-3#. The patients who will be found unsuitable for brachytherapy will be kept under observation. Week 12: After treatment completion, response assessment will be done using following parameters: • Pain assessment using numerical pain rating scale on 0-10 • Vaginal bleeding- yes/no • Vaginal discharge- yes/ no • Analgesic use- WHO ladder and dosing • QOL QC30, QLQC15 Pall, QLQC Cervix 24 • Disease response • Acute toxicity. Follow up: Patients follow up will be utilizing standard of care imaging and lab investigations used for the patients. Patients will be evaluated every 3 months for the study duration.
  Interventions: Radiation: Short course palliative radiation.

INTERVENTIONS:
Radiation: Short course palliative radiation. — Week 1: Patients in the experimental arm will be treated with short course radiotherapy (25Gy/5#). The dose fractionation of 25 Gy in 5# over a week will be used. Week 4: Patients who have almost complete clinical response will be evaluated for brachytherapy will receive the appropriate brachytherapy procedure depending on the tumor response to a dose of 6-8Gy x 2-3#. The patients who will be found unsuitable for brachytherapy will be kept under observation. Week 12: After treatment completion, response assessment will be done using following parameters: • Pain assessment using numerical pain rating scale on 0-10 • Vaginal bleeding- yes/no • Vaginal discharge- yes/ no • Analgesic use- WHO ladder and dosing • QOL QC30, QLQC15 Pall, QLQC Cervix 24 • Disease response • Acute toxicity. Follow up: Patients follow up will be utilizing standard of care imaging and lab investigations used for the patients. Patients will be evaluated every 3 months for the study duration.
  Arms: Arm B or Experimental Arm-Short course palliative radiation.
Radiation: Long course palliative treatment. — Week1: All the patients will receive external sitting of radiation treatment, first fraction of 10 Gy. Week4: All the patients will receive external sitting of radiation treatment, second fraction of 10 Gy. Week7: Patients who have almost complete clinical response will be evaluated for brachytherapy will receive the appropriate brachytherapy procedure depending on the tumor response to a dose of 6-8Gy x 2-3#.The patients who will be found unsuitable for brachytherapy will receive another sitting of external radiation, third fraction of 10 Gy. Week 12: After treatment completion response assessment will be done using following parameters: • Pain assessment using numerical pain rating scale on 0-10 • Vaginal bleeding- yes/ no • Vaginal discharge- yes/no • Analgesic use- WHO ladder and dosing • QOL QC30, QLQC15 Pall, QLQC Cervix 24 • Disease response • Acute toxicity
  Arms: Arm A Or Control Arm- Long course palliative treatment.

SUMMARY:
The present study is proposed to compare a rapid fractionation schedule of 1 week compared to a protracted schedule of 6-8 weeks for palliation for locally advanced cervical cancer.

DETAILED DESCRIPTION:
This is a prospective randomised open label Phase III study. This study is is proposed to compare a rapid fractionation schedule of 1 week compared to a protracted schedule of 6-8 weeks for palliation for locally advanced cervical cancer. The primary objective of the study is pain relief in the experimental arm as compared to the control arm from treatment until 12 weeks from start of radiotherapy. Patients with locally advanced cervical cancer (Stage III B-IV A) deemed unsuitable for full course radical pelvic radiotherapy or chemoradiation, patients whose anticipated survival is less than 12 months will be included in the study. Patients with distant metastasis and those with retroviral disease will be excluded from the study. The patients will be randomised in one of the two groups:

Arm A : Control Arm - Long Course Palliative Radiation: Week 1: All the patients will receive external sitting of radiation treatment, first fraction of 10 Gy. Week 4: All the patients will receive external sitting of radiation treatment, second fraction of 10 Gy. Week 7: Patients who have almost complete clinical response will be evaluated for brachytherapy will receive the appropriate brachytherapy procedure depending on the tumor response to a dose of 6-8Gy x 2-3#.The patients which will be found unsuitable for brachytherapy will receive another sitting of external radiation, third fraction of 10 Gy. Week 12: After treatment completion response assessment will be done using following parameters: • Pain assessment using numerical pain rating scale on 0-10 • Vaginal bleeding- yes/ no • Vaginal discharge- yes/no • Analgesic use- WHO ladder and dosing • QOL QC30, QLQC15 Pall, QLQC Cervix 24 • Disease response • Acute toxicity.

Arm B: Experimental arm- Short Course Palliative radiation. Week 1: Patients will be treated with short course radiotherapy (25Gy/5#). The dose fractionation of 25 Gy in 5# over a week will be used. Week 4: Patients who have almost complete clinical response will be evaluated for brachytherapy will receive the appropriate brachytherapy procedure depending on the tumor response to a dose of 6-8Gy x 2-3#. The patients who will be found unsuitable for brachytherapy will be kept under observation. Week 12: After treatment completion response assessment will be done using following parameters: • Pain assessment using numerical pain rating scale on 0-10 • Vaginal bleeding- yes/no • Vaginal discharge- yes/ no • Analgesic use- WHO ladder and dosing • QOL QC30, QLQC15 Pall, QLQC Cervix 24 • Disease response • Acute toxicity. Follow up: Patients follow up will be utilizing standard of care imaging and lab investigations used for the patients. Patients will be evaluated every 3 months for the study duration.There is no potential direct benefit to the study participants. However the aim is to use the available information to evolve treatment in future. The variables to be estimated are pain relief, disease related symptoms relief, CTCAE Toxicity, Quality of Life,overall survival and compliance to therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Locally advanced cervical cancer (Stage IIIB-IVA) deemed unsuitable for full course radical pelvic radiotherapy or chemoradiation due to the following reasons:

   * Very large volume hard fixed disease infiltrating pelvic wall muscles and ligaments on clinical examination also classified clinically as "frozen pelvis" wherein curative intent treatment is not envisaged or feasible.
   * Fistulous communication between tumour growth and rectum and bladder >2x2 cm in size (as judged by cystoscopy for bladder infiltration or clinical or proctosigmoidoscopy examination for rectal/sigmoid infiltration) wherein radical intent treatment is not intended or feasible and patient is not a candidate for pelvic exenteration.
   * Deranged renal parameters as measured by Serum Creatinine >3 mg/dl wherein diversion nephrostomy is not planned by the multidisciplinary team due to anticipated poor clinical outcomes.Furthermore concurrence for palliative intent radiotherapy should be corroborated by 2 staff radiation oncologists.
2. Moderate to Severe Pain on Numerical Rating Score (Score 4 or higher).
3. Anticipated survival < 12 months.
4. Patients with stage IVB with local disease extent as described in section 1 but systemic chemotherapy is not possible either due to deranged renal function or anticipated poor tolerance.

Exclusion Criteria:

1. Patients with distant metastasis needing upfront systemic therapy.
2. Presence of retroviral disease
3. Non-compliant for follow up.
4. Expected survival <3 months.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is about cervical cancer.
Enrollment: 230 (Estimated)
Dates: Start 2020-06-19 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Pain Relief (Numerical pain rating scale will be used) | 1 week, 4 week, 7 week, 12 weeks
  Pain relief in the experimental arm as compared to the control arm from treatment until 12 weeks from start of radiotherapy will be assessed.
  Pain relief will be assessed at 12 weeks from start of radiotherapy. (Pain has been chosen as the primary endpoint as it is the primary complaint in almost 2/3 rd of patients. Numerical pain rating scale has been chosen for objective pain assessment as it is easy to use and has been proven to be a reliable tool in multiple studies.
  Pain score will be documented on 11-scale numerical pain rating scale (NRS) and qualified into one of the following categories:
  i)Pain score of 0-3- No to mild pain ii)Pain score 4-7- Moderate pain iii)Pain score >7- Severe pain

SECONDARY OUTCOMES:
Pain Relief (Numerical pain rating scale will be used) | 6 months, 9 months, 12 months
  Pain relief at 6, 9 and 12 month of follow up.
  Pain score will be documented on 11-scale numerical pain rating scale (NRS) and qualified into one of the following categories:
  i) Pain score of 0-3- No to mild pain ii) Pain score 4-7- Moderate pain iii) Pain score >7- Severe pain
Presence or absence of vaginal bleeding and/or discharge and relief in vaginal bleeding (as reported by the patient) | 1 week,4 week,7week,12 weeks
  Complete relief in vaginal bleeding and non-infectious discharge will be documented at 12 weeks from start of RT as reported by the patient. Although vaginal bleeding and discharge are also major presenting complaints, there is no standardized objective scale or criteria for measuring these in cancer patients.
  Vaginal discharge if present will be qualified as infectious or non-infectious. Infectious vaginal discharge will warrant antibiotic treatment.
Change in use of analgesics (WHO ladder) | 12 weeks, 3 month, 9 month, 12 month
  Change in use of analgesics by either dose adjustment or stepping up/down on the WHO ladder at 12 weeks.This will also be recorded at each clinical follow up.
Compliance to therapy | 7 week,12 week, 3 month, 9 month, 12 month
  Response of local disease will be assessed clinically at end of treatment and on every follow up. Response to RT will be determined on follow-up at 7 and 12 weeks in both the arms and phone call interviews when necessary for completeness in patients with poor compliance to follow up.
Quality of Life using EORTC QLQC30 questionnaires | At start of radiotherapy, 12 week and at 3, 6, 9 & 12 months follow up.
  Quality of Life using EORTC QLQC 30 questionnaire (European Organisation for Research & Treatment of Cancer - Quality of Life Questionnaire of Cancer patients) will be evaluated at start of radiotherapy and at week 12, 3 month, 6 month, 9 month,12 months follow up.
  Scale- Not at all-1 , A little Bit-2, Quite a bit-3, very much-4.
  1 will be considered as better outcome & 4 will be considered as worst outcome.
Quality of Life using EORTC QLQC-15 Pall questionnaires | At start of radiotherapy, 12 week and at 3, 6, 9 & 12 months follow up.
  Quality of Life using EORTC QLQC-15 Pall (European Organisation for Research & Treatment of Cancer - Quality of Life Questionnaire in Palliative Cancer care patients) will be evaluated at start of radiotherapy and at week 12, 3 month, 6 month, 9 month,12 months follow up.
  Scale- Not at all-1 , A little Bit-2, Quite a bit-3, very much-4.
  1 will be considered as better outcome & 4 will be considered as worst outcome.
Quality of Life using Cx-24 questionnaires | At start of radiotherapy, 12 week and at 3, 6, 9 & 12 months follow up.
  Quality of Life using Cx-24 questionnaires (European Organisation for Research & Treatment of Cancer - Quality of Life Questionnaire of Cervical cancer patients) will be evaluated at start of radiotherapy and at week 12, 3 month, 6 month, 9 month,12 months follow up.
  Scale- Not at all-1 , A little Bit-2, Quite a bit-3, very much-4.
  1 will be considered as better outcome & 4 will be considered as worst outcome.
Acute gastrointestinal and genitourinary toxicities | Within 90 days of Radiotherapy
  Acute gastrointestinal and genitourinary toxicities using CTCAE ver4.0 grading will be measured within 90 days of Radiotherapy.
Late gastrointestinal and genitourinary toxicities | After 90 days of Radiotherapy
  Late gastrointestinal and genitourinary toxicities using CTCAE 4.0 grading will be measured after 90 days of Radiotherapy.
Overall survival, defined as time from randomization until death due to any cause. | 1 year
  Overall survival, defined as time from randomization until death due to any cause.
Patterns of terminal event (Due to local relapse or Distant Metastasis) | By telephonic interview of the relatives at 3, 6, 9 or 12 months, as applicable
  Events leading to death will be determined by telephonic interview of the relatives at 3, 6, 9 or 12 months, as applicable to find out the terminal cause of death.

CONTACTS AND LOCATIONS:
Overall Officials: Supriya Sastri, Principal Investigator — Tata Memorial Hospital
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided